CLINICAL TRIAL: NCT00950521
Title: Phase II Study of Autologous Peripheral Blood CD34 Stem Cell Implantation in Chronic Stroke Patients
Brief Title: Efficacy Study of CD34 Stem Cell in Chronic Stroke Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Shinn-Zong Lin M.D., Ph.D., Professor of Neurosurgery, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMR-96-IRB-145; DOH Approval No:098004365
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Stroke; Middle Cerebral Artery Infarction
Keywords: Stroke; Stem Cell; Cell Therapy; CD34 Stem cell; Peripheral blood Stem cell
MeSH Terms: conditions — Stroke; Infarction, Middle Cerebral Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PBSC Treatment (Active Comparator): Patients in PBSC treatment will receive brain implant of autologous peripheral blood stem cell(CD34+) plus convention stroke treatment that include rehabilitation and antiplatelet medication
  Interventions: Procedure: Intercerebral implantation of Autulogous Stem Cells
- Control (Active Comparator): Control group receive conventional stroke treatment that include rehabilitation and antiplatelet medication
  Interventions: Drug: convention therapy

INTERVENTIONS:
Procedure: Intercerebral implantation of Autulogous Stem Cells — 2-8 millions Stem cell per patients plus convention therapy
  Other Names: PBSC; CD34 Stem Cell
  Arms: PBSC Treatment
Drug: convention therapy — antiplatelet
  Arms: Control

SUMMARY:
The objective of the study is to determine the efficacy of brain transplants of CD34+ stem cells obtained from peripheral blood of patients in the treatment of chronic stroke patients.

DETAILED DESCRIPTION:
30 patients are divided into 2 groups, one treatment group and one control group.Treatment group will be implanted with peripheral blood stem cell and receive convention stroke therapy ,and control group only receive convention stroke therapy. We expect that transplantation of the peripheral blood CD34+ cells has the potential of significant benefit to neurological recovery. In a previous phase I clinical trial, we have shown that transplantation of CD34+ cells obtained from the peripheral blood of the chronic stroke patients was safe and beneficial for neurological recovery. We expect this trial can further prove the efficacy of this treatment method.

ELIGIBILITY:
Inclusion Criteria:

* aged 35-70 chronic stroke adult patient,
* with stroke history of more than 6 months, less than 60 months，
* with stable hemiplegia condition, and
* NIHSS (NIH Stroke Scale) score is between 9-20.

Exclusion Criteria:

* patients aged less than 35 or more than 70,
* hemorrhage stroke or MRI show the occlusion is not in the middle cerebral artery territory，NIHSS is not in the range of 9-20,
* pregnant women,
* impaired liver function, abnormal blood coagulation, AIDS, combine other tumor or special condition.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
NIH-stroke scale (NIHSS) | 1, 2, 4, 12 weeks, and confirmed at 6 and 12 months

SECONDARY OUTCOMES:
European stroke scale (ESS) | 1, 2, 4, 12 weeks, and confirmed at 6 and 12 months
European stroke motor subscale (EMS) | 1, 2, 4, 12 weeks, and confirmed at 6 and 12 months
Barthel index and Mini-Mental State Examination (MMSE) | 1, 2, 4, 12 weeks, and confirmed at 6 and 12 months
Magnetic resonance imaging (MRI) and computed tomography (CT) scans | 1, 2, 4, 12 weeks, and confirmed at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shinn-Zong Lin, MD, DMSci, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Mackie AR, Losordo DW. CD34-positive stem cells: in the treatment of heart and vascular disease in human beings. Tex Heart Inst J. 2011;38(5):474-85. PMID 22163120